CLINICAL TRIAL: NCT06133374
Title: Concordance of Molecular Classification Based on Fine Needle Biopsy (FNB) and Surgical Samples
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: Qualisure Diagnostics Inc. (Unknown); Alberta Health services (Other)
Responsible Party: Sponsor
Other Study IDs: HREBA.CC-23-0001
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Papillary Thyroid Cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fine needle biopsy sample, frozen tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to determine whether results from a fine needle biopsy are the same as results from a larger sample that is acquired from the surgical pathology using the Thyroid GuidePx® test in patients with papillary thyroid carcinoma.

DETAILED DESCRIPTION:
Thyroid cancer is the 8th most common cancer, and incidence has been increasing. Papillary thyroid carcinoma (PTC) accounts for most thyroid cancers. Treatment decisions related to PTC depend on the doctor's estimate on whether the cancer is aggressive or not. Current methods for distinguishing aggressive tumors from less aggressive tumors rely on clinical factors as well as factors related to the final pathology (after the tumor has been removed). Ideally, the information required to make decisions would be available prior to surgery, so that surgical decisions can be made.

A new test is being developed to determine molecular features of a PTC and to estimate the risk of cancer recurrence after surgery. Thyroid GuidePx® provides unique information that may inform doctors' decisions. The greatest potential for Thyroid GuidePx® to impact on clinical care is if it can be performed prior to surgery on a fine needle biopsy (FNB). If Thyroid GuidePx® could be done on an FNB, it would inform surgeons on the type of surgery that would be most appropriate for an individual.

A recent feasibility study consisting of 12 patients with PTC demonstrated that performing the Thyroid GuidePx® assay on FNBs is feasible. However, reliance on a limited FNB for molecular disease characterization implies that the sample is representative of the entirety of the tumor. Genomic and transcriptomic heterogeneity has been described in primary tumors and metastases. Therefore, it will be important to document the concordance between samples acquired by FNB and surgical samples. The goal of this study is to determine whether the more limited sample from an FNB is sufficiently representative of the larger tumor to determine a valid molecular classification using the Thyroid GuidePx® test in patients with PTC.

Participants will be invited to participate if they have a preoperative tissue diagnosis of PTC (Bethesda VI) or suspicious for PTC (Bethesda V), and they are eligible for partial or total thyroidectomy. During surgery, when the thyroid gland and the tumor are exposed, the surgeon will perform an FNB of the dominant tumor (ie: the lesion identified preoperatively), under direct vision. The cellular material from the FNB will be sent for processing. Separate surgical samples will be processed and examined. This will follow routine specimen processing protocols and will not interfere with standard methods of pathologic diagnosis. Tissue will be released for research only once sufficient tissue is taken for diagnostic and clinical use. RNASeq for Thyroid GuidePx® for both FNB and surgical samples will be performed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* A diagnosis of papillary thyroid cancer based on a fine needle biopsy (FNB) interpreted as a Bethesda V or VI cytology
* A diagnosis of Atypia of Undetermined Significance (AUS) or Follicular Lesion of Undetermined Significance (FLUS) interpreted as Bethesda III or IV cytology (indeterminate nodule) ThyroSpec positive for BRAFV600E, TERT, rearrangements in BRAF, RET, NTRK1, NTRK3, RAS + TERT, RAS + EIF1AX, AKT1, PI3CA, CTNNB1, EGFR, rearrangements in ALK
* Tumor size > 1 cm in maximal diameter on imaging prior to surgery
* The patient is an operative candidate
* The patient has provided consent

Exclusion Criteria:

* History of radiation to the neck for situations such as medical radiation, radiation exposure in a work environment (nuclear power plant/reactor), or radiation exposure through release of radioactive materials into the nearby environment from a nuclear power plant/reactor.
* Unable or unwilling to have a fine needle biopsy
* Unwilling to undergo thyroidectomy
* Final pathology does not demonstrate papillary thyroid cancer
* Cases where there is no clear dominant nodule
* Cases where there are multiple nodules that preclude sampling of a defined nodule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a preoperative tissue diagnosis of PTC (Bethesda VI) or suspicious for PTC (Bethesda V) or a tissue diagnosis of Undetermined Significance (AUS) or Follicular Lesion of Undetermined Significance (FLUS) interpreted as Bethesda III or IV cytology (indeterminate nodule) ThyroSpec positive for BRAFV600E, TERT, rearrangements in BRAF, RET, NTRK1, NTRK3, RAS + TERT, RAS + EIF1AX, AKT1, PI3CA, CTNNB1, EGFR, rearrangements in ALK, eligible for partial or total thyroidectomy
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Concordance between Thyroid GuidePx® molecular classifications acquired from FNAs and matched frozen surgical samples | December 1, 2025
  The molecular class assignment (Type 1, Type 2 and Type 3), based on the pattern of expression of prognostic genes, will be compared between samples obtained by FNB and matched frozen surgical specimens. The significance of concordance between the two sample types will be determined using the kappa statistic.

SECONDARY OUTCOMES:
The technical success rate in completing a valid Thyroid GuidePx® using FNB and FFPE surgical samples | December 1, 2025
  Sufficient RNA of good quality to perform the test
The recurrence outcomes using the ATA risk stratification system vs. patients classified by Thyroid GuidePx® using surgical samples | May 1, 2028
  Biochemical and structural recurrence
The test performance of Thyroid GuidePx® as a prognostic test (FNB and surgical samples) in comparison to ATA Risk Stratification. | May 1, 2028
  Specificity, sensitivity, AUROC, positive predictive value, and negative predictive value,

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Yeo, MD, Principal Investigator — Alberta Health services
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davies L, Morris LG, Haymart M, Chen AY, Goldenberg D, Morris J, Ogilvie JB, Terris DJ, Netterville J, Wong RJ, Randolph G; AACE Endocrine Surgery Scientific Committee. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY DISEASE STATE CLINICAL REVIEW: THE INCREASING INCIDENCE OF THYROID CANCER. Endocr Pract. 2015 Jun;21(6):686-96. doi: 10.4158/EP14466.DSCR. PMID 26135963
- [Background] Sciuto R, Romano L, Rea S, Marandino F, Sperduti I, Maini CL. Natural history and clinical outcome of differentiated thyroid carcinoma: a retrospective analysis of 1503 patients treated at a single institution. Ann Oncol. 2009 Oct;20(10):1728-35. doi: 10.1093/annonc/mdp050. PMID 19773250
- [Background] Pacini F, Castagna MG. Approach to and treatment of differentiated thyroid carcinoma. Med Clin North Am. 2012 Mar;96(2):369-83. doi: 10.1016/j.mcna.2012.01.002. Epub 2012 Feb 10. PMID 22443981
- [Background] Tuttle RM, Tala H, Shah J, Leboeuf R, Ghossein R, Gonen M, Brokhin M, Omry G, Fagin JA, Shaha A. Estimating risk of recurrence in differentiated thyroid cancer after total thyroidectomy and radioactive iodine remnant ablation: using response to therapy variables to modify the initial risk estimates predicted by the new American Thyroid Association staging system. Thyroid. 2010 Dec;20(12):1341-9. doi: 10.1089/thy.2010.0178. Epub 2010 Oct 29. PMID 21034228
- [Background] Castagna MG, Maino F, Cipri C, Belardini V, Theodoropoulou A, Cevenini G, Pacini F. Delayed risk stratification, to include the response to initial treatment (surgery and radioiodine ablation), has better outcome predictivity in differentiated thyroid cancer patients. Eur J Endocrinol. 2011 Sep;165(3):441-6. doi: 10.1530/EJE-11-0466. Epub 2011 Jul 12. PMID 21750043
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Background] Cheng SP, Chien MN, Wang TY, Lee JJ, Lee CC, Liu CL. Reconsideration of tumor size threshold for total thyroidectomy in differentiated thyroid cancer. Surgery. 2018 Sep;164(3):504-510. doi: 10.1016/j.surg.2018.04.019. Epub 2018 May 26. PMID 29843911
- [Background] Dhir M, McCoy KL, Ohori NP, Adkisson CD, LeBeau SO, Carty SE, Yip L. Correct extent of thyroidectomy is poorly predicted preoperatively by the guidelines of the American Thyroid Association for low and intermediate risk thyroid cancers. Surgery. 2018 Jan;163(1):81-87. doi: 10.1016/j.surg.2017.04.029. Epub 2017 Nov 8. PMID 29128185
- [Background] Lang BH, Shek TW, Wan KY. The significance of unrecognized histological high-risk features on response to therapy in papillary thyroid carcinoma measuring 1-4 cm: implications for completion thyroidectomy following lobectomy. Clin Endocrinol (Oxf). 2017 Feb;86(2):236-242. doi: 10.1111/cen.13165. Epub 2016 Sep 1. PMID 27467318
- [Background] Kluijfhout WP, Pasternak JD, Lim J, Kwon JS, Vriens MR, Clark OH, Shen WT, Gosnell JE, Suh I, Duh QY. Frequency of High-Risk Characteristics Requiring Total Thyroidectomy for 1-4 cm Well-Differentiated Thyroid Cancer. Thyroid. 2016 Jun;26(6):820-4. doi: 10.1089/thy.2015.0495. Epub 2016 May 20. PMID 27083216
- [Background] Murthy SP, Balasubramanian D, Subramaniam N, Nair G, Babu MJC, Rathod PV, Thankappan K, Iyer S, Vijayan SN, Prasad C, Nair V. Prevalence of adverse pathological features in 1 to 4 cm low-risk differentiated thyroid carcinoma. Head Neck. 2018 Jun;40(6):1214-1218. doi: 10.1002/hed.25099. Epub 2018 Feb 8. PMID 29417654
- [Background] Craig SJ, Bysice AM, Nakoneshny SC, Pasieka JL, Chandarana SP. The Identification of Intraoperative Risk Factors Can Reduce, but Not Exclude, the Need for Completion Thyroidectomy in Low-Risk Papillary Thyroid Cancer Patients. Thyroid. 2020 Feb;30(2):222-228. doi: 10.1089/thy.2019.0274. Epub 2020 Jan 9. PMID 31813323
- [Background] Cancer Genome Atlas Research Network. Integrated genomic characterization of papillary thyroid carcinoma. Cell. 2014 Oct 23;159(3):676-90. doi: 10.1016/j.cell.2014.09.050. PMID 25417114
- [Background] Craig S, Stretch C, Farshidfar F, Sheka D, Alabi N, Siddiqui A, Kopciuk K, Park YJ, Khalil M, Khan F, Harvey A, Bathe OF. A clinically useful and biologically informative genomic classifier for papillary thyroid cancer. Front Endocrinol (Lausanne). 2023 Sep 12;14:1220617. doi: 10.3389/fendo.2023.1220617. eCollection 2023. PMID 37772080
- [Background] Rubino C, de Vathaire F, Dottorini ME, Hall P, Schvartz C, Couette JE, Dondon MG, Abbas MT, Langlois C, Schlumberger M. Second primary malignancies in thyroid cancer patients. Br J Cancer. 2003 Nov 3;89(9):1638-44. doi: 10.1038/sj.bjc.6601319. PMID 14583762
- [Background] Pitoia F, Jerkovich F, Urciuoli C, Schmidt A, Abelleira E, Bueno F, Cross G, Tuttle RM. Implementing the Modified 2009 American Thyroid Association Risk Stratification System in Thyroid Cancer Patients with Low and Intermediate Risk of Recurrence. Thyroid. 2015 Nov;25(11):1235-42. doi: 10.1089/thy.2015.0121. Epub 2015 Aug 6. PMID 26132983
- [Background] Zhou H, Mody DR, Smith D, Lloyd MB, Kemppainen J, Houghton J, Wylie D, Szafranska-Schwarzbach AE, Takei H. FNA needle rinses preserved in Cytolyt are acceptable specimen type for mutation testing of thyroid nodules. J Am Soc Cytopathol. 2015 May-Jun;4(3):128-135. doi: 10.1016/j.jasc.2015.01.001. Epub 2015 Jan 9. PMID 31051693
- [Background] Fuller MY, Mody D, Hull A, Pepper K, Hendrickson H, Olsen R. Next-Generation Sequencing Identifies Gene Mutations That Are Predictive of Malignancy in Residual Needle Rinses Collected From Fine-Needle Aspirations of Thyroid Nodules. Arch Pathol Lab Med. 2018 Feb;142(2):178-183. doi: 10.5858/arpa.2017-0136-OA. Epub 2017 May 24. PMID 28537807
- [Background] Chen T, Gilfix BM, Rivera J, Sadeghi N, Richardson K, Hier MP, Forest VI, Fishman D, Caglar D, Pusztaszeri M, Mitmaker EJ, Payne RJ. The Role of the ThyroSeq v3 Molecular Test in the Surgical Management of Thyroid Nodules in the Canadian Public Health Care Setting. Thyroid. 2020 Sep;30(9):1280-1287. doi: 10.1089/thy.2019.0539. Epub 2020 May 5. PMID 32242511
- [Background] Eszlinger M, Bohme K, Ullmann M, Gorke F, Siebolts U, Neumann A, Franzius C, Adam S, Molwitz T, Landvogt C, Amro B, Hach A, Feldmann B, Graf D, Wefer A, Niemann R, Bullmann C, Klaushenke G, Santen R, Tonshoff G, Ivancevic V, Kogler A, Bell E, Lorenz B, Kluge G, Hartenstein C, Ruschenburg I, Paschke R. Evaluation of a Two-Year Routine Application of Molecular Testing of Thyroid Fine-Needle Aspirations Using a Seven-Gene Panel in a Primary Referral Setting in Germany. Thyroid. 2017 Mar;27(3):402-411. doi: 10.1089/thy.2016.0445. Epub 2017 Feb 7. PMID 28071986
- [Background] Titov S, Demenkov PS, Lukyanov SA, Sergiyko SV, Katanyan GA, Veryaskina YA, Ivanov MK. Preoperative detection of malignancy in fine-needle aspiration cytology (FNAC) smears with indeterminate cytology (Bethesda III, IV) by a combined molecular classifier. J Clin Pathol. 2020 Nov;73(11):722-727. doi: 10.1136/jclinpath-2020-206445. Epub 2020 Mar 25. PMID 32213552
- [Background] Gonzalez HE, Martinez JR, Vargas-Salas S, Solar A, Veliz L, Cruz F, Arias T, Loyola S, Horvath E, Tala H, Traipe E, Meneses M, Marin L, Wohllk N, Diaz RE, Veliz J, Pineda P, Arroyo P, Mena N, Bracamonte M, Miranda G, Bruce E, Urra S. A 10-Gene Classifier for Indeterminate Thyroid Nodules: Development and Multicenter Accuracy Study. Thyroid. 2017 Aug;27(8):1058-1067. doi: 10.1089/thy.2017.0067. Epub 2017 Jul 11. PMID 28521616
- [Background] Le Pennec S, Konopka T, Gacquer D, Fimereli D, Tarabichi M, Tomas G, Savagner F, Decaussin-Petrucci M, Tresallet C, Andry G, Larsimont D, Detours V, Maenhaut C. Intratumor heterogeneity and clonal evolution in an aggressive papillary thyroid cancer and matched metastases. Endocr Relat Cancer. 2015 Apr;22(2):205-16. doi: 10.1530/ERC-14-0351. Epub 2015 Feb 17. PMID 25691441
- [Background] Kamarudin AN, Cox T, Kolamunnage-Dona R. Time-dependent ROC curve analysis in medical research: current methods and applications. BMC Med Res Methodol. 2017 Apr 7;17(1):53. doi: 10.1186/s12874-017-0332-6. PMID 28388943
- [Background] Flack V, Afifi A, Lachenbruch P, Schouten H. Sample size determinations for the two rater kappa statistic. Psychometrika. 1988;53(3):321-5.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT06133374/Prot_SAP_002.pdf
  • Informed Consent Form (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT06133374/ICF_001.pdf